CLINICAL TRIAL: NCT06426472
Title: The Effect of Web-Based Support Program on Psychosocial Health Status in Women With Unsuccessful IVF Experience
Brief Title: An Intervention on Psychosocial Health in Women With Unsuccessful IVF Experience
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Elif Balkan, PhD Student, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: EBIstanbulUC; 1649B032306898 (Other Grant/Funding Number: TUBITAK)
Record Dates: First submitted 2024-05-14; First posted 2024-05-23 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Infertility; Failed in Vitro Fertilisation
Keywords: infertility; web-based; support; psychosocial health
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Interventional group which will be given the web-based fertility support
  Interventions: Other: Web-based support program
- Control (No Intervention): Control group will not be given any intervention

INTERVENTIONS:
Other: Web-based support program — Web-based support program for infertile women with failed IVF experience
  Arms: Intervention

SUMMARY:
The goal of this interventional study is to learn if web-based support program can improve the psychosocial health status in women with unsuccessful IVF experience. The main questions it aims to answer are:

Does web-based support decrease the depressive symptoms, anxiety and infertility-related stress? Does web-based support decrease the hopelessness? Does web-based support increase the coping skills with infertility-related stress?

Researchers will compare this intervention to a control group to see if web-based support program improves psychosocial health.

Participants will:

Use the web-based support intervention for 5 weeks or have no intervention. Complete the surveys on the website before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Having at least three repeated unsuccessful IVF experiences,
2. Maximum one month has passed since the negative IVF experience,
3. Participating in the study voluntarily,
4. Being able to read, understand and communicate in Turkish.

Exclusion criteria

1. Not having access to the internet/not knowing how to use it,
2. Having any psychiatric disease/being in the 'severe depression' grade as a result of the Beck Depression Inventory,
3. Having at least one living child.

Exclusion criteria from the study in the stages after including the study:

1. Spontaneous pregnancy occurring,
2. Starting a new treatment cycle,
3. Not continuing to monitor the modules on the website.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Depression (Beck Depression Inventory) | 24 months
  Beck Depression Inventory (BDI) will be used to evaluate the participants' anxiety outcome. This inventory, whose validity and reliability in Turkish was studied by Hisli (1989), consists of a total of 21 items and four interpreted sub-dimensions. The scoring of the scale is a four-point Likert type (0 = positive statements about depression; 3 = negative statements about depression). The total score that can be obtained from the scale varies between 0-63; 0-9 points indicate minimal depression, 10-16 points indicate mild depression, 17-29 points indicate moderate depression, and 30-63 points indicate severe depression.
Infertility-related stress (The Infertility Stress Scale) | 24 months
  The Infertility Stress Scale will be used to assess participants' infertility-related stress. Schmidt (2006) developed this scale in 1996. In our country, the validity and reliability of the scale was studied by Şahin Yılmaz (2012). This scale is a scale with a total of 14 items consisting of three sub-dimensions and answers are given in a Lykert type. Calculations per subdimensions requires a special formula for each subdimension. An increase in score is interpreted as an increase in stress.
Coping Skills with Infertility Stress (Coping with Infertility Stress Scale) | 24 months
  Coping with Infertility Stress Scale: Developed by Schmidt (2006) in 1996. In our country, the validity and reliability of the scale was studied by Şahin Yılmaz (2012). This scale is a scale with a total of 19 items consisting of four sub-dimensions.
  e Active-Struggle Coping, Passive-Struggle Coping, Passive-Ignoring Coping and Meaning-Based Coping Method. Each subscale score can be calculated seperately.

SECONDARY OUTCOMES:
Hopelessness | 24 months
  Beck Hopelessness Scale: Beck et al. (1974) to measure the individual's negative expectations for the future. Although the Turkish adaptation of this scale was made by Seber (1993), Durak (1994) examined the validity, reliability and factor structure of the scale in more detail. The scale consists of a total of 20 questions and the answers are given as true/false. The scale consists of three subscales: feelings about the future, loss of motivation, and expectations about the future. 1 point for incorrect answers to items 1-3-5-6-8-10-13-15 and 19, and 1 point for correct answers to items 2-4-7-9-11-14-16-17-18 and 20. and a total score between 0 and 20 can be obtained from the scale. The "arithmetic sum" found by calculation is accepted as the "despair score". The scale does not have a cut-off score; as the scores obtained from the scale increase, it is interpreted that the individual's level of hopelessness also increases.
Effect of the Web-based study program | 24 months
  Web-Based Psychosocial Support Evaluation Form: It is an 8-question form created by researchers to evaluate opinions about the psychosocial support initiative applied to the web-based support program.
  System Usability Scale: The Turkish validity and reliability of the scale developed by Brooke (1996) was tested by Demirkol and Şeneler (2018). "The scale consisting of ten items is a five-point Likert type (1=Strongly Disagree, 2=Disagree, 3=Undecided, 4=Agree, 5=Strongly Agree)." Items numbered 1, 3, 5, 7, 9 in the scale are scored positively, and items numbered 2, 4, 6, 8, 10 are reverse scored because they contain negative expressions. The answer "I strongly disagree" is calculated as "0" and the answer "I strongly agree" is calculated as 4 points. To obtain the total score, the score from each item is multiplied by 2.5 to obtain a score ranging from 0 to 100. A score between 65-70 is sufficient to show that the website is usable.